CLINICAL TRIAL: NCT00244582
Title: Direct Convection-Enhanced Delivery of Glucocerebrosidase for the Treatment of Type 2 (Acute Neuronopathic) Gaucher Disease
Brief Title: Convection-Enhanced Delivery of Glucocerebrosidase to Treat Type 2 Gaucher Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060007; 06-N-0007
Record Dates: First submitted 2005-10-26; First posted 2005-10-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-11-03

CONDITIONS: Type 2 Gaucher Disease
Keywords: Central Nervous System; Enzyme Replacement Therapy; Convection; Gaucher Disease; Neuronopathic Gaucher Disease; Type 2 Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

SUMMARY:
This study will use an experimental method of delivering the enzyme glucocerebrosidase directly into the brain of a patient with Gaucher disease to treat disease symptoms. Patients with Gaucher disease have insufficient levels of glucocerebrosidase. As a result, substances normally broken down by this enzyme accumulate in the body, causing damage to the brain and other organs. Symptoms of Gaucher disease outside the brain can be treated by infusing the missing enzyme intravenously (IV, through a vein). However, IV infusions do not help the neurologic symptoms of the disease, because the enzyme cannot get into the brain. This study will use a new technique called convection-enhanced delivery to try to introduce glucocerebrosidase directly into the brain.

This single-patient study includes an 8-month-old male with Type 2 Gaucher disease with progressive neurological decline.

In preparation for the enzyme infusion, the patient will have a complete physical examination, including a detailed neurological examination, and blood and urine tests. On the day of surgery, the child will be placed under general anesthesia for magnetic resonance imaging (MRI) of the brain. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. For this procedure, the child lies on a table that is moved into the scanner (a narrow cylinder), wearing earplugs to protect his hearing from the loud knocking and thumping sounds that occur during the scanning process. He will then be brought to the operating room for the infusion procedure, as follows:

An incision will be made in the scalp and a small hole drilled through the skull. Then, a small tube (cannula) will be positioned through the hole into the target area in the brain. Once the tip of the cannula is in place, it will be connected with tubing to a syringe filled with glucocerebrosidase in saline (salt water). The child will then have a second MRI scan to make sure the cannula is placed correctly and to monitor delivery of the glucocerebrosidase to the brain. The child will be monitored closely with MRI scans every 30 to 60 minutes during the infusion to look for fluid in the brain and determine the extent of the enzyme perfusion. The infusion will last no longer than 6 hours and will be stopped when the full dose of enzyme has been delivered. The cannula will be removed and the scalp incision closed. The child will stay in the hospital for observation from 4 to 10 days, with at least 24 hours in the intensive care unit and 3 to 7 days in the pediatric unit.

The child will be seen in the clinic two weeks after discharge and then once a month for 3 months to evaluate any possible effects of the surgery. These follow-up visits include a repeat MRI scan and neurological examination. After the first 3 months, visits may be less frequent.

If the child continues to have symptoms during the course of follow-up or his neurologic status worsens, additional enzyme infusions will be offered, possibly including treatment of the brainstem. If the child gains no benefit after three infusions have been performed, no additional infusions will be offered. If there appears to be any neurological benefit, additional infusions may be offered.

DETAILED DESCRIPTION:
Objective. To overcome the previous delivery limitations and to provide enzyme to the deficient sites in the central nervous system (CNS) of a Type 2 Gaucher disease patient, we will investigate the use of convection-enhanced delivery (CED) to perfuse specific sites within the CNS with glucocerebrosidase in an effort to ameliorate that patient's neurologic symptomatology and prolong his life.

Study population. This is a single patient study that includes a male infant (8 months of age) with Type 2 Gaucher disease that has been diagnosed by clinical, laboratory and genetic testing. The natural history of acute neuronopathic (Type 2) Gaucher disease is progressive neurological decline that is rapidly fatal.

Design. We propose using CED of glucocerebrosidase to the CNS to treat the neurologic signs and symptoms in this Type 2 Gaucher patient. Regions of infusion within the CNS will be targeted based on neurologic findings.

Outcome measures. Detailed clinical and neurologic examinations will be performed pre- (3 days before infusion) and post-infusion (1, 14, 30, and 90 days after infusion then every 3 months until study completion) to determine stabilization or improvement in neurologic signs and symptoms. Survival will also be used to determine the efficacy of this treatment.

ELIGIBILITY:
* INCLUSION CRITERIA

The patient is eligible because he has Type 2 Gaucher disease.

EXCLUSION CRITERIA

The patient may not be eligible to receive CED of glucocerebrosidase if he:

1. Is not healthy enough to undergo surgery or general anesthesia.
2. Has an uncorrectable bleeding disorder.
3. Is not able to undergo magnetic resonance (MR)-imaging.

Max Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1
Dates: Start 2005-10-22; Study Completion 2006-11-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Barton NW, Brady RO, Dambrosia JM, Di Bisceglie AM, Doppelt SH, Hill SC, Mankin HJ, Murray GJ, Parker RI, Argoff CE, et al. Replacement therapy for inherited enzyme deficiency--macrophage-targeted glucocerebrosidase for Gaucher's disease. N Engl J Med. 1991 May 23;324(21):1464-70. doi: 10.1056/NEJM199105233242104. PMID 2023606